CLINICAL TRIAL: NCT05276180
Title: Evaluation of Implementation and Effectiveness of a Multifactorial Intervention Strategy for Safe Patient Handling and Movement in the Healthcare Sector - A Cluster Randomized Controlled Trial
Brief Title: Evaluation of Interventions for Safe Patient Handling and Movement in the Healthcare Sector
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Östergötland (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Charlotte Wåhlin, Associate professor, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Dnr: 190144 (AFA insurance)
Record Dates: First submitted 2022-02-11; First posted 2022-03-11 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Occupational Health
Keywords: healthcare; Safety climate; patient handling; risk assessment; guideline; education; occupational safety and health; healthcare workers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A) Multifactorial intervention strategy (Experimental): Experimental: Multifactorial intervention strategy for safe patient handling and movement (PHM) - Arm A The multifactorial intervention strategy for care units randomized to Arm A includes: 1) Swedish guideline for PHM and digital introduction for using the guideline (two workshops for manager and implementation team) 2) Training modules (theoretical and practical - one session) 3) Risk assessment with TilThermometer (four times) and 4) Fall risk assessment using Downton Fall Risk Index (DFRI) or existing fall risk assessment instrument at the care unit (all patients) and 5) Work environment mapping with Structured Multidisciplinary Work Environment Survey (SMET) including active/personal feedback
  Interventions: Other: Arm A) Multifactorial intervention strategy
- Arm B) Single intervention strategy (Active Comparator): No further interventions other than access to the Swedish guideline for patient handling and movement and the results from the SMET questionnaire will be presented to the manager. Arm B will be assigned an external facilitator who provides information, is present at the start-up meeting and will be the contact person during the study period. No further support will be given to the care units in arm B.
  Interventions: Other: Arm B) Single intervention strategy

INTERVENTIONS:
Other: Arm A) Multifactorial intervention strategy — Implementation of the multifactorial intervention strategy will be supported by the following components:
  1) An implementation team at each intervention unit consisting of 5-6 HCWs is responsible for informing and engaging all HCWs at the unit. For implementing the various components of the strategy. They will have the role of planning regular workplace meetings. 2) One or two internal facilitators will be the link between the external facilitator and the care unit. The internal facilitator will give support with material, information and will be able to ask questions of the external facilitator.
  3) External facilitator will ensure that the implementation process works according to plan. The research team will present the results of SMET to the implementation team.
  4) The research group will be project leaders and support the external facilitators. They will provide workshops and will also be responsible for data collection.
  Arms: Arm A) Multifactorial intervention strategy
Other: Arm B) Single intervention strategy — No further interventions other than access to the Swedish guideline for patient handling and movement and the results from the SMET questionnaire will be presented to the manager. Arm B will be assigned an external facilitator who provides information, is present at the start-up meeting and will be the contact person during the study period. No further support will be given to the care units in arm B.
  Arms: Arm B) Single intervention strategy

SUMMARY:
There are several situations in the workplace in which both healthcare workers and patients are at risk of injury. Frequent patient transfers, heavy lifting and patient mobilization are proven risk factors for musculoskeletal disorders among healthcare workers. Falls and patient transfers are frequently reported causes of patient injuries. Swedish occupational safety and health legislation and the Patient Safety Act require employers to provide good, safe care and to conduct risk assessments to prevent risks and injuries in the healthcare sector. It has been suggested that a combination of workplace interventions is needed to facilitate safe patient handling and movement and to prevent musculoskeletal disorders and injuries among healthcare workers and patients.

The main aim of the cluster randomized and controlled trial (RCT) is to evaluate a multifactorial intervention strategy that includes risk assessment instruments as well as guidelines and training. This strategy will be compared with a single intervention strategy for safe patient handling and movement in workplaces in the Swedish regional and municipal healthcare system. All healthcare workers in the care units recruited to this RCT will be invited to participate. The study will evaluate the intervention strategies with regard to primary outcome measures given equal priority according to a hybrid 2 design of the RCT. These are: 1) the implementation process (acceptability, appropriateness and feasibility), here called the implementation outcome, and 2) the effect of the applied strategies (measured with regard to the workplace safety climate and additional questions about safety for patient handling and movement), here called intervention effectiveness.

This RCT is part of the Swedish Patient and Workers Safety Study (PAWSS). The aim of the PAWSS project is to contribute to a regional and municipal healthcare that is evidence-based and organized for both patient safety and a safe working environment for healthcare workers. The long-term goal is to facilitate safe patient handling and movement practices which prevent both care injuries and work injuries.

DETAILED DESCRIPTION:
There are several risk factors in the healthcare environment which lead to work-related injuries among healthcare workers (HCWs) and harmful incidents for patients. In previous research on patient injuries and HCW incidents and injuries, the results indicate that both patient safety and occupational safety for HCWs are insufficient. Common occupational injuries among healthcare professionals were those caused by sharp objects or needles; exposure to infection; injuries that occur in threatening and violent situations; and injuries that occur during patient handling and movement (PHM). Musculoskeletal disorders that occur in connection with PHM are one of the most common injuries. The starting point for a safe environment and a strengthened safety climate is that the employer, together with HCWs and safety representatives, regularly examines and assesses the risks that exist in the daily work routine and provides proper interventions to create a good work environment. A Swedish national guideline for safe PHM is being developed by the research group in 2022. It will be used in the present study in combination with the participating care units' existing patient safety work and work environment policies. There is a need to increase the use of risk assessment and promote intervention strategies in the healthcare sector that can facilitate safe PHM. A recent systematic review by Wåhlin and co-authors shows that a number of work interventions can be effective for safe PHM. These include providing equipment and training workers, since it can increase their use of equipment. Training workers to be peer coaches is also associated with fewer injuries. Other effective strategies for safe PHM are participatory ergonomics and management engagement with staff. There is great interest among employers, HCWs and other stakeholders in providing effective interventions that can promote health, prevent musculoskeletal disorders among HCWs and prevent patient injuries. At present, however, there is a lack of knowledge regarding how risk assessments and comprehensive interventions need to be tailored to be effective and how learning for safe PHM should be designed to be perceived as useful in a clinical setting.

The main aim of the cluster randomized controlled trial (RCT) is to implement and evaluate a multifactorial intervention strategy for safe PHM and compare it with a single intervention strategy. The trial will be carried out in workplaces in the regional and municipal healthcare system. The study will evaluate the two strategies with regard to the implementation outcome (acceptability, appropriateness and feasibility) and the intervention effectiveness of the applied strategies (safety climate in relation to aspects of patient handling and movement). With a hybrid 2 design, implementation outcome and intervention effectiveness are given equal priority. The hypothesis in this study is that care units that receive the multifactorial intervention strategy develop a stronger and more appropriate safety climate with specific focus on PHM compared with units that receive a single intervention strategy. The hypothesis is tested by performing a randomized controlled study with pre- and post-measurements among care units in regions and municipalities in Sweden.

Method and material: The study for the implementation of intervention strategies for safe PHM will be carried out in least twelve units in regional and municipal health care in Sweden. The study design is a cluster randomized controlled study in which participating care units are randomized into two randomization arms: Arm A or Arm B. At least six units (Arm A) will receive a multifactorial intervention strategy and at least six will receive a single intervention strategy (Arm B).

The multifactorial intervention strategy for care units randomized to Arm A consists of: 1) a Swedish guideline for PHM and a digital introduction to using the guideline, 2) training modules (theoretical and practical), 3) risk assessment with TilThermometer, 4) a fall risk assessment using Downton Fall Risk Index or a fall risk assessment instrument in use at the care unit, and 5) work environment mapping with the Structured Multidisciplinary Work Environment Survey (SMET). The intervention strategies for safe PHM will be used at the participating units over a 4-month period. They will however be encouraged by the project coordinators to continue to promote safe PHM until the 12-month follow up questionnaire is answered by HCWs at the participating units.

An implementation team will be created at each intervention unit. The team will consist of 5-6 people, including the manager, a range of healthcare professions and safety representatives. The intervention units (Arm A) will be offered support from the project during the implementation process (four months) to create good conditions for implementation (facilitator). The results from the SMET questionnaire will be presented to the implementation team along with interviews with the manager and discussions about the systematic work environment management. The results from SMET will also be presented to the process team after four months.

Training will be offered to all HCWs. One session of practical training for safe PHM and theoretical education will be offered online. Participating units in Arm A will be able to discuss the Swedish guideline for PHM at two workshops. Here, participants will discuss themes and the guidelines' recommendations. The process team will formulate a number of problem areas they want to work with in the workplace using a participatory approach. The TilThermometer will be used for risk assessment four times during the implementation period.

Arm A will be encouraged to involve their occupational health care services and have an active collaboration during the 4-month implementation period.

The active comparator, healthcare units randomized to Arm B, will receive the single intervention strategy. The participants will receive an online introduction to the Swedish guideline for PHM. They will be encourage to apply the content of the guideline in order to promote safe PHM at their care unit. The results from the SMET questionnaire will be presented to the manager.

Recruitment of units: To recruit care units, information will be distibuted to workplaces in the Swedish regional and municipal healthcare system, via contact persons such as HR managers and managers. The research project will have the support of the reference group that has been put together for the project and consists of various stakeholders. Information will also be disseminated via advertisements in trade union newspapers and the project will be highlighted by means of newspaper interviews. Several communication channels will also be used to recruit units.

Information about the study and what participation entails will be sent out to managers and given at workplace meetings or the equivalent. The manager will sign a written consent before the care unit's participation in the study.

Prior to start-up, staff from the research group will give further information about the study and the procedure for collecting consent to each group. The HCWs will be invited to participate in the study via the care unit's common email groups or equivalent. They will also be given further information at workplace meetings or equivalent. All participants will be given the opportunity to ask questions and get more information.

Each unit that has agreed to participate in the study will have a start-up meeting to introduce the strategy that the unit will work with, Arm A or Arm B.

Inclusion Criteria: In regional healthcare: inpatient units/wards. In municipal healthcare: nursing homes for the elderly. Where a recruited clinic has several care units, they will be counted as one cluster. Exclusion Criteria: Units providing home nursing outpatient clinics; and clinics providing paediatric, emergency and psychiatric care.

A power calculation has been made where estimation of number of cluster and participants in each cluster was calculated. A power level of 0.8 (80%) and alpha 0.05 is used. The calculation resulted in at least six units/clusters for each arm with minimum of 15 participants in each unit/cluster.

The care units will be randomized by a computer-generated randomization-list to either Arm A or Arm B after stratification in blocks by the size of the care unit and type of organization. A care unit is defined as one which has one manager who is responsible for all employees (HCWs) at the unit.

Outcome and data collection HCWs working in care units which are participating in the study will be able to read the consent and send in their own consent. In doing so they agree to participate in the study and answer three questionnaires. Data collection will be performed at baseline and at 4-month and 12-month follow ups. In the case of participating care units (Arm A), information about the interview study will be disseminated during the implementation period by means of workplace meetings, email and the project's website. Prior to participating in individual interviews and focus group discussions, participants will sign a consent form, either digitally or in paper format.

This study will evaluate a multifactorial versus a single strategy for safe PHM. It will look at the implementation process (acceptability, appropriateness and feasibility) and the effect of the applied strategies (safety climate in relation to aspects of patient handling and movements). These are the primary outcomes which are refered to as implementation outcome and intervention effectiveness. The following contextual factors will be collected from each participating care unit: number of risk assessments the previous year; number of managers; number of HCWs; number of admissions care recipients / places; care burden; number of inpatients; completed work environment training previous year; current work environment policy; completed training in PHM.

At the start of the study (baseline), the participating HCWs and managers (Arm A and Arm B) will be asked to answer a questionnaire. The questionnaire will be sent out again after completion of the implementation (four months) and at follow-up after 12 months. The participating units will be encouraged to continue on their own to promote safe patient handling and movement and to work according to the multifactorial intervention strategy or the single intervention strategy. Background data will be included in the baseline questionnaire, such as age, education, gender, working full time/part time, overtime, profession, years of experience in the profession and current workplace. Contextual factors and changes (mediators) at the unit that may affect the implementation process will be collected. A study specific logbook will be used. Contextual factors can be for example staff turnover, work organizational changes, interventions for occupational safety and health, unforeseen events and so on.

Primary outcome, implementation outcome: the implementation outcome (acceptability, appropriateness and feasibility) will be measured by a standardized questionnaire to evaluate the usefulness/benefit of the multifactorial intervention strategy. For the evaluation of the implementation process, a mixed design will be used that includes both quantitative and qualitative data. Primary outcome, intervention effectiveness: The intervention effectiveness will be measured with regard to the safety climate in the workplace and an additional question about safety for patient handling and movement.

All data will be documented via digital collection platforms and collected at baseline and at 4-month and 12-month follow ups. All data in the research project will be collected in a digital data collection tool. Interviews will be collected after the 4-month implementation period.

All collected data will be stored so that no unauthorized persons have access to it. Results and characteristics of participating individuals will be presented at group level or in such a way that individuals cannot be identified.

ELIGIBILITY:
Inclusion Criteria:

* In regional healthcare: inpatient units/wards.
* In municipal healthcare: nursing homes for the elderly.
* Where a recruited clinic has several care units, they will be counted as one cluster.

Exclusion Criteria:

* Units providing home nursing outpatient clinics
* Clinics at hospitals providing paediatric care
* Clinics at hospital providing emergency care
* Clinics at hospital providing psychiatric care.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2060 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Intervention effectiveness - Change in 50 items across 7 safety climate dimensions and 14 items of safety for patient handling and movement | Change from Baseline at 4 months follow up and 12 months follow up.
  NOSACQ-50 The questionnaire consists of 50 items across 7 safety climate dimensions (Management safety priority, commitment, and competence, Management safety empowerment, Management safety justice, Workers' safety commitment, Workers' safety priority and risk non-acceptance, Safety communication, learning, and trust in co-workers safety competence, Trust in the efficacy of safety systems) in the workplace, additional 14 specific research-based questions to evaluate the safety climate for patient handling and movement will be used. Involving dimensions of using equipment, other aspects of safety, performing risk assessment and co-production between caregivers and patients.
  The questionnaire use a score with the scale 1-4, where 1 is labeled as "Not correct at all" and 4 is labeled as "Completely correct".
  A score of more than 3.30 indicates a good level of safety climate.
Acceptability - Implementation outcome | 4 months follow up
  Acceptability of Intervention Measure (AIM), 4 questions with five units on a scale (1-5), 1 is labeled "disagree" and 5 is labeled "fully agree". Higher scores indicates a better outcome.
Acceptability - Implementation outcome | 12 months follow up
  Acceptability of Intervention Measure (AIM), 4 questions with five units on a scale (1-5), 1 is labeled "disagree" and 5 is labeled "fully agree". Higher scores indicates a better outcome.
Appropriateness - Implementation outcome | 4 months follow up
  Intervention Appropriateness Measure (IAM), 4 questions with five units on a scale (1-5), 1 is labeled "disagree" and 5 is labeled "fully agree". Higher scores indicates a better outcome.
Appropriateness - Implementation outcome | 12 months follow up
  Intervention Appropriateness Measure (IAM), 4 questions with five units on a scale (1-5), 1 is labeled "disagree" and 5 is labeled "fully agree". Higher scores indicates a better outcome.
Feasability - Implementation outcome | 4 months follow up
  Feasibility of Intervention Measure (FIM), 4 questions with five units on a scale (1-5), 1 is labeled "disagree" and 5 is labeled "fully agree". Higher scores indicates a better outcome.
Feasability - Implementation outcome | 12 months follow up
  Feasibility of Intervention Measure (FIM), 4 questions with five units on a scale (1-5), 1 is labeled "disagree" and 5 is labeled "fully agree". Higher scores indicates a better outcome.

SECONDARY OUTCOMES:
Evaluation of the work environment | Change from baseline at four months follow up and twelve months follow up.
  The Structured Multidisciplinary Work Evaluation Tool (SMET) will be used. The questionnaire asks about physically, environmentally and psychosocially demanding work items (30 items). A scale of 1-10 is used in the questionnaire, 1 is labeled "Not at all" and 10 is labeled "Highly".
Global Health | Change from baseline at 4 months follow up and 12 months follow up.
  General self-reported health obtained by the question: "In general, would you say your health is…?", with five anchor points ranging between excellent and poor.
Work strain | Change from Baseline at 4 months follow up and 12 months follow up.
  Borg-CR 10 in general, specific for patient handling and movement, and for muscle strength.
  A sacle 0-10 is used. 0 is labeled "No one at all" and 10 is labeled "Extremely strong".
Work performance - work ability | Change from baseline at 4 months follow up and 12 months follow up.
  WAI (Work Ability Index) single item, physical and mental demands in work, sick-leave, sickness work capacity
Perceived work environment problems | Change from baseline at 4 months follow up and 12 months follow up.
  Employees are asked whether they have experienced any work environment problems in the previous seven days. Work environment problems are defined as any physical, psychological or social problems that resulted from the work environment. Response options are yes/no
Work environment related production loss | Change from baseline at 4 months follow up and 12 months follow up.
  During the past 7 days, how much did your work environment-related problems affect your performance at work? A scale 0 - 10 is used, 0 is labeled " Work environment problems have not affected my work performance" and 10 is labeled "Work environment problems completely prevented me from working". A higher score indicates a worse outcome.
Sickness presence | Change from baseline at 4 months follow up and 12 months follow up.
  During the past 7 days, have you had a health related problem/illness but still chosen to go to work? Yes or No. If yes, a scale from 0-10 is used, where 0 is labeled " Health problems have not affected my work performance" and 10 is labeled as "Health problems completely prevented me from working"
Sickness influence on ability to work | Change from baseline at 4 months follow up and 12 months follow up.
  Is your disorder or injury affecting your ability to work? Range from no problem to being sickness absent.
Sickness absence | Change from baseline at 4 months follow up and 12 months follow up.
  How many days have you been absent from work in the last 12 months because of sickness or injury? A scale from 1 - 5 is used, where 1 is labeled as "100-365 days" and 5 is labeled as "no days", a higher score indicates a better outcome
Work related musculoskeletal disorders (WMSD) | Change from baseline at 4 months follow up and 12 months follow up.
  Pain and symptoms of the musculoskeletal system. Questions about the presence of pain and symptoms of the neck, shoulders, elbows, wrists/hands, upper back, lower back, one hip or both, one knee or both, and one ankle or both. Yes and no is used for WMSD has been present during last 12 months and 7 days. If yes, a scale wiht 1-10 is used for assesing the intensity, 1 is labeled "no problems" and 10 is labeled "Problems as difficult as they can ever be".
Fit for work - physical strength | Change from baseline at 4 months follow up and 12 months follow up.
  Individual physical strength: How do you evaluate your muscle strength in comparison to others? A scale 0-10 is used, 0 is labeled "Much weaker" and 10 is labeled "Much stronger".
  It is not better or worse whether you score high or low.
Daily physcial acitivty | Change from baseline at 4 months follow up and 12 months follow up.
  How much "everyday exercise" have you received in the last 12 months by, for example, walking or cycling to work, school, bus stop, shop, etc. or by going out with the dog, shoveling snow, working in the garden or the like?¨ A scale with 4 item is used, from "not at all" to "daily activity".
Physcial exercise the last 12 months | Change from baseline at 4 months follow up and 12 months follow up.
  To what extent have you in the last 12 months engaged in any voluntary exercise / sports / outdoor activity in addition to the everyday exercise that you have stated above? A scale with 5 items is used, from "Very low physical activity" to "I regularly devoted myself to hard exercise or competition where the physical effort was great"
Strenuous physical activity | Change from baseline at 4 months follow up and 12 months follow up.
  How much time do you spend a regular week doing physical exercise, which makes you breathless, such as running, gymnastics, ball sports? A scale with 6 items is used, from "0 minutes/no time at all" to "More than 120 minutes"
Time of daily physical activity | Change from baseline at 4 months follow up and 12 months follow up.
  How much time do you spend a regular week doing everyday exercise, such as walking, cycling, gardening? Add up all the time (at least 10 minutes at a time) A scale with 7 items is used, from "0 minutes/no time at all" to "More than 300 minutes"
Fidelity | Through study completion, an average of 4 months
  To measure fidelity (to which extent the intervention in ARM A has been followed as intended) a study specific logbook will be used. The logbook contains the 5 steps in the intervention strategy; 1) Number of workshops being performed by the manager and implementation team 2) Number of healthcare workers attending training modules 3) Number of risk assessment with TilThermometer 4) Percentage of fall risk assessment of all patients during the implementation period 5) Performed SMET with active feedback
Managers and implementation team members' experiences with the intervention strategy and implementation process | After the 4 months study period.
  This data will be collected using semi-structured interviews.
Healthcare workers' experiences of the intervention strategy and implementation process | After the 4 months study period.
  This data will be collected through focus-group discussions.

CONTACTS AND LOCATIONS:
Overall Officials: charlotte Wåhlin, Ass. prof., Principal Investigator — Arbets- och miljömedicin, Region Östergötland/Linköpings Universitet
Locations (1):
- Depatment of Occupational Medicine, Linköping, Ösgtergötland, Sweden

IPD SHARING:
Plan to Share IPD: Yes
As a government agency, LiU come under the Public Access to Information and Secrecy Act .Research data can therefore be requested to be disclosed.
  Project research data can be made accessible online or following a request submitted to the principal investigator.
  Possible restrictions that can affect the possibilities of making research data accessible.
  Responsibility for long-term preservation stays with the principal investigator after the completion of the project
  The research project uses Region Östergötlands secure drives to store research data on. It will also be stored in the Archives of Region Östergötland.
  For datasets to be accessible in the future, they need to be saved in future-proofed formats. Ahead of a possible publication of data files, they will be future-proofed.
  A data management plan is available on request from the principal investigator.
Time Frame: Data will become available after scientific publication. Estimated earliest at 2026.
Access Criteria: Data can be requested from the principal investigator.

REFERENCES:
- [Background] Strid EN, Wahlin C, Ros A, Kvarnstrom S. Health care workers' experiences of workplace incidents that posed a risk of patient and worker injury: a critical incident technique analysis. BMC Health Serv Res. 2021 May 27;21(1):511. doi: 10.1186/s12913-021-06517-x. PMID 34044852
- [Background] Wahlin C, Stigmar K, Nilsing Strid E. A systematic review of work interventions to promote safe patient handling and movement in the healthcare sector. Int J Occup Saf Ergon. 2022 Dec;28(4):2520-2532. doi: 10.1080/10803548.2021.2007660. Epub 2021 Dec 19. PMID 34789085
- [Derived] Wahlin C, Sandqvist J, Enthoven P, Buck S, Karlsson N, Strid EN. Perceived health, musculoskeletal disorders, work conditions and safety climate in relation to patient handling and movement - a multicentre cross-sectional study at healthcare workplaces. BMC Musculoskelet Disord. 2025 Nov 14;26(1):1048. doi: 10.1186/s12891-025-09330-3. PMID 41239349
- [Derived] Wahlin C, Buck S, Sandqvist J, Enthoven P, Fock J, Andreassen M, Strid EN. Evaluation of the implementation and effectiveness of a multifactorial intervention strategy for safe patient handling and movement in the healthcare sector: a study protocol of a cluster randomised controlled trial. BMJ Open. 2023 Feb 3;13(2):e067693. doi: 10.1136/bmjopen-2022-067693. PMID 36737081